CLINICAL TRIAL: NCT04860700
Title: A Phase 2 Study of Anlotinib in Patients With Metastatic Pheochromocytoma or Paraganglioma
Brief Title: The Efficacy and Safety of Anlotinib in Patients With Metastatic Pheochromocytoma or Paraganglioma
Status: Completed | Phase: Phase 2 | Type: Interventional
Sponsor: Peking Union Medical College Hospital (Other)
Responsible Party: Sponsor
Allocation: Not Applicable | Model: Single Group | Masking: None | Purpose: Treatment
Other Study IDs: PUMCHMPPGL
Record Dates: First submitted 2021-04-22; First posted 2021-04-27 (Actual); Last update posted 2024-06-12 (Actual); Status verified 2023-04

CONDITIONS: Malignant Adrenal Gland Pheochromocytoma; Malignant Paraganglioma; Pheochromocytoma, Metastatic; Paraganglioma, Malignant; Paraganglioma, Extra-Adrenal
Keywords: pheochromocytoma; paraganglioma; Metastatic; inoperable
MeSH Terms: conditions — Paraganglioma, Extra-Adrenal; Pheochromocytoma; Neoplasm Metastasis; Paraganglioma | interventions — anlotinib

STUDY DESIGN:
Oversight: Data Monitoring Committee: Yes | FDA-regulated Drug: No | FDA-regulated Device: No

ARMS (1):
- anlotinib hydrochloride (Experimental): Patients receive anlotinib hydrochloride 12mg orally once daily on days 1-14. Courses repeat every 21 days in the absence of disease progression or unacceptable toxicity.
  Interventions: Drug: anlotinib hydrochloride

INTERVENTIONS:
Drug: anlotinib hydrochloride — Patients receive anlotinib hydrochloride 12mg orally once daily on days 1-14. Courses repeat every 21 days in the absence of disease progression or unacceptable toxicity.
  Other Names: anlotinib

SUMMARY:
This phase II trial studies how well anlotinib hydrochloride works in treating patients with metastatic pheochromocytoma or paraganglioma. Anlotinib hydrochloride may stop the growth of tumor cells by blocking some of the enzymes needed for cell growth and by blocking blood flow to the tumor.

DETAILED DESCRIPTION:
PRIMARY OBJECTIVES:

To determine the anti-tumor activity of anlotinib hydrochloride (Objective Response rate,ORR) in patients with metastatic pheochromocytomas or paragangliomas.

SECONDARY OBJECTIVES:

I. To assess safety profile of anlotinib. II. To assess progression-free survival time. III. To assess disease control rate.

OUTLINE:

Patients receive anlotinib hydrochloride 12mg orally once daily on days 1-14. Courses repeat every 21 days in the absence of disease progression or unacceptable toxicity.

Patients undergo urine and blood sample collection, imaging examinations at baseline and periodically during study.

After completion of study therapy, patients are followed up every 3-6 months.

ELIGIBILITY:
Inclusion Criteria:

1. Provide written informed consent.
2. Willing to return to enrolling institution for follow-up.
3. Eastern Cooperative Oncology Group (ECOG) performance status 0, 1, or 2.
4. Life expectancy > 3 months.
5. Patients diagnosis with metastatic pheochromocytoma or paraganglioma that is unresectable.
6. Laboratory requirements:

1）Absolute granulocyte count (AGC) greater than 1.5 x 109/L; 2）Platelet count greater than 80 x 109/L; 3) Hemoglobin greater than 90g/L; 4) Serum bilirubin less than 1.5 x upper limit of normal (ULN); 5)Serum aspartate aminotransferase (AST) and alanine aminotransferase (ALT) less than 2.5 x ULN; 6) Serum creatinine less than 1.5 x ULN or creatinine clearance (CCr)≥60ml/min; 7.Doppler ultrasound assessment: left ventricular ejection fraction (LVEF) ≥ lower limit of normal value (50%).

Exclusion Criteria:

1. Any of the following:Pregnant women,Nursing women,Men or women of childbearing potential who are unwilling to employ adequate contraception.
2. Patients who have previously used other anti-vascular targeted drugs, such as sunitinib, bevacizumab, endurance, etc.
3. Chemotherapy/systemic therapy, radiotherapy, immunotherapy or surgery within 4 weeks prior to kinase inhibitor therapy.
4. Patients with another primary malignancy within 5 years prior to starting study drug, with the exception of adequately treated in-situ carcinoma of the uterine cervix, or skin cancer (such as basal cell carcinoma, squamous cell carcinoma, or non-melanomatous skin cancer).
5. Those who have multiple factors that affect oral medications (such as inability to swallow, chronic diarrhea, intestinal obstruction, etc.).
6. Patients with known untreated brain metastases are excluded. Patients having a history of brain metastasis that have been previously irradiated or resected greater than 2 months prior to enrollment and are clinically and radiographically stable will be considered for enrollment. Patients with brain metastases with symptoms or symptom control for less than 2 months.
7. Active or uncontrolled intercurrent illness including, but not limited to 1)Patients with unsatisfactory blood pressure control (systolic blood pressure ≥150 mmHg, diastolic blood pressure ≥100 mmHg); 2) Patients with uncontrolled myocardial ischemia or myocardial infarction, arrhythmia (including QTC≥480ms), and uncontrolled congestive heart failure，grade ≥2（New York Heart Association ）; 3) ongoing or active infection; 4) Liver cirrhosis, decompensated liver disease, active hepatitis or chronic hepatitis require antiviral treatment; 5) Renal failure requires hemodialysis or peritoneal dialysis; 6) Have a history of immunodeficiency, including HIV or other acquired or congenital immunodeficiency diseases, or a history of organ transplantation; 7) Diabetes is poorly controlled (fasting blood glucose (FBG)> 10mmol/L); 8) Urine routines suggest that urine protein is ≥++, and the 24-hour urine protein content is confirmed to be greater than 1.0 g; 9) Patients who have seizures and need treatment;
8. Any of the following conditions =< 6 months prior to registration: Cerebrovascular accident (CVA) or transient ischemic attack (TIA); Serious or unstable cardiac arrhythmia; Pulmonary embolism, untreated deep venous thrombosis (DVT).
9. Received major surgical treatment, open biopsy or obvious traumatic injury within 28 days before enrollment.
10. Those who have a history of psychotropic drug abuse and cannot be quit or have mental disorders.
11. Imaging shows that the tumor has invaded important blood vessels or the investigator judges that the tumor is very likely to invade important blood vessels and cause fatal bleeding during the follow-up study.
12. Regardless of the severity, patients with any signs of bleeding or medical history; within 4 weeks before enrollment, patients with any bleeding or bleeding event ≥ CTCAE grade 3, unhealed wounds, ulcers or fractures.
13. Participated in other clinical trials within 4 weeks.
14. Patients are using drugs that interact with Anlotinib.

Ages: 18 Years to 75 Years | Sex: All | Healthy Volunteers: Yes
Age Groups: Adult, Older Adult
Enrollment: 27 (Actual)
Dates: Start 2021-04-30 (Actual); Primary Completion 2023-10-17 (Actual); Study Completion 2023-10-17 (Actual)

PRIMARY OUTCOMES:
Objective Response rate RECIST Using Version 1.1 | minimum of 4 cycles
  Defined for all patients whose tumor met the criteria of Complete Response (CR)and Partial Response (PR)

SECONDARY OUTCOMES:
Disease Control Rate | minimum of 4 cycles
  Defined for all patients whose tumor met the criteria of CR or PR or stable disease(SD)

OTHER OUTCOMES:
Progression-free Survival Time | minimum of 4 cycles
  PFS is defined as the time from the first day of treatment to the first documented disease progression per RECIST 1.1 criteria and the Kaplan-Meier curve. Changes in only the largest diameter (unidimensional measurement) of the tumor lesions are used in the RECIST criteria.
Incidence of adverse events assessed by Common Terminology Criteria for Adverse safety profile of anlotinib | minimum of 4 cycles
  Incidence of adverse events assessed by Common Terminology Criteria for Adverse Events version 4.0

CONTACTS AND LOCATIONS:
Overall Officials: Anli Tong, Principal Investigator — Peking Union Medical College Hospital
Locations (1):
- Peking Union Medical College Hospital, Beijing, Beijing Municipality, China

IPD SHARING:
Plan to Share IPD: No